CLINICAL TRIAL: NCT02487745
Title: The Long-Term Treatment of Drug Addiction and Unemployment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00046990; R01DA037314-01A1 (NIH)
Record Dates: First submitted 2015-06-19; First posted 2015-07-01 (Estimated); Results first posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-07

CONDITIONS: Substance Abuse, Intravenous
Keywords: Cocaine; Methadone; Employment; Opioids
MeSH Terms: conditions — Substance Abuse, Intravenous | interventions — Palliative Care; Myo-Inositol-1-Phosphate Synthase; Employment, Supported

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IPS Only (Active Comparator): IPS Only participants will receive the Individual Placement and Support (IPS) supported employment.
  Interventions: Behavioral: Individual Placement and Support (IPS) supported employment
- IPS Plus Wage Supplement (Experimental): IPS Plus Abstinence-Contingent Wage Supplement participants will receive the Individual Placement and Support (IPS) supported employment intervention and abstinence-contingent wage supplements.
  Interventions: Behavioral: Abstinence-contingent wage supplements; Behavioral: Individual Placement and Support (IPS) supported employment

INTERVENTIONS:
Behavioral: Abstinence-contingent wage supplements — Before obtaining competitive employment, participants will be able to earn wage supplements for attending two individual placement and support (IPS) supported employment sessions per week, and for completing specific tasks prescribed by IPS including developing a worker profile, applying for appropriate jobs, and completing job interviews. Once a participant becomes employed, participants will be able to earn up to $5 per hour for every hour worked in a competitive job up to 40 hours per week verified by pay stubs. To maintain long-term drug abstinence, participants will be required to provide urine samples to earn the maximum in wage supplements.
  Arms: IPS Plus Wage Supplement
Behavioral: Individual Placement and Support (IPS) supported employment — Individual Placement and Support (IPS) supported employment involves rapid job search, promotes competitive employment, considers the participant's preferences, and provides job supports and benefits counseling. An employment specialist will establish relationships will potential employers and work with participants to identify potential jobs, prepare applications, and to apply for positions.

SUMMARY:
The purpose of this clinical trial is to evaluate the effectiveness and economic benefits of a Wage Supplement Model of arranging long-term exposure to employment-based abstinence reinforcement.

DETAILED DESCRIPTION:
Drug addiction is as a chronic relapsing disorder. High magnitude and long-duration voucher-based abstinence reinforcement is one of the most effective treatments for drug addiction and can maintain drug abstinence over extended periods of time, but practical methods of implementing these interventions are needed. Workplaces could be ideal and practical vehicles for arranging and maintaining abstinence reinforcement over long time periods. The investigator's research on a model Therapeutic Workplace has shown that employment-based abstinence reinforcement, in which participants must provide drug-free urine samples to maintain maximum pay, can maintain drug abstinence. Now what is needed is the development of effective and economically sound methods to arrange long-term exposure to employment-based abstinence reinforcement. The present study will evaluate the effectiveness and economic benefits of a Wage Supplement Model of arranging long-term exposure to employment-based abstinence reinforcement. Under this model, successful Therapeutic Workplace participants are offered abstinence-contingent wage supplements if they obtain and maintain competitive employment. Governments have used wage supplements effectively to increase employment in welfare recipients. The Wage Supplement Model harnesses the power of wage supplements to promote employment, while simultaneously using the wage supplements to reinforce drug abstinence. The intervention will combine the Therapeutic Workplace, Individual Placement and Support (IPS) supported employment, and abstinence-contingent wage supplements. IPS is a supported employment intervention that has been proven effective in promoting employment in adults with severe mental illness. Under this model, participants will be exposed to the Therapeutic Workplace to initiate drug abstinence and establish job skills. To promote employment and prevent relapse to drug use, participants will receive IPS Plus Abstinence-Contingent Wage Supplements. A randomized trial will evaluate the effectiveness and economic benefits of the Abstinence-Contingent Wage Supplement Model in promoting employment and sustaining abstinence in heroin users. Participants will be enrolled in the Therapeutic Workplace for 3 months and then randomly assigned to an IPS Only group or an IPS Plus Abstinence-Contingent Wage Supplement group for one year. IPS Only participants will receive the IPS intervention. IPS Plus Abstinence-Contingent Wage Supplement participants will receive the IPS intervention and abstinence-contingent wage supplements. Drug use while participants are employed in community jobs will be monitored by American Substance Abuse Professionals, Inc. (ASAP®), a leading provider of workplace substance abuse services in the U.S. This novel intervention could be an effective and economically sound way to promote long-term abstinence and employment.

ELIGIBILITY:
Inclusion Criteria:

* report heroin use

Exclusion Criteria:

* report current suicidal or homicidal ideation;
* have a severe psychiatric disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-11; Primary Completion 2019-09 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Silverman, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Center for Learning and Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The data will be published in a peer-reviewed journal.

REFERENCES:
- [Derived] Holtyn AF, Toegel F, Subramaniam S, Jarvis BP, Leoutsakos JM, Fingerhood M, Silverman K. Abstinence-contingent wage supplements to promote drug abstinence and employment: a randomised controlled trial. J Epidemiol Community Health. 2020 May;74(5):445-452. doi: 10.1136/jech-2020-213761. Epub 2020 Feb 21. PMID 32086373

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled in a 3-month abstinence initiation phase (Phase 1) prior to random assignment.
Period: Overall Study
Arm/Group | IPS Only | IPS Plus Wage Supplement
Started | 47 | 44
Completed | 47 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IPS Only | IPS Plus Wage Supplement | Total
Number analyzed (Participants) | 47 | 44 | 91
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 44 | 89
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 27 | 23 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 46 | 38 | 84
  Unknown or Not Reported | 1 | 4 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 28 | 51
  White | 22 | 14 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47 | 44 | 91

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Opiate- and Cocaine-negative Urine Samples
Description: (# opiate- and cocaine-negative urine samples/divided by possible #) x 100
Time Frame: 1 year
Population: Intent-to-treat
Measure: Mean (Full Range); unit: percentage of urine samples
Arm/Group | IPS Only | IPS Plus Wage Supplement
Number analyzed (Participants) | 47 | 44
percentage of urine samples | 44.9 [0 to 100] | 64.6 [0 to 100]
Statistical Analysis 1: Comparison: IPS Only vs IPS Plus Wage Supplement; Test type: Superiority; p = .05, Regression, Logistic; Odds Ratio (OR) = 2.29

2. Primary Outcome: The Percentage of Participants Who Are Employed
Description: (# participants employed /divided by total # of participants) x 100
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Arm/Group | IPS Only | IPS Plus Wage Supplement
Number analyzed (Participants) | 47 | 44
percentage of participants | 27.7 | 59.1
Statistical Analysis 1: Comparison: IPS Only vs IPS Plus Wage Supplement; Test type: Superiority; p = .05, Regression, Logistic; Odds Ratio (OR) = 3.88

3. Secondary Outcome: The Percentage of Participants Who Report Injecting Drugs
Description: (# participants reporting injecting drugs /divided by total # of participants) x 100
Time Frame: 1 year
Reporting Status: Not Posted

4. Secondary Outcome: The Percentage of Participants Who Report Trading Unprotected Sex for Drugs or Money
Description: (# participants reporting trading unprotected sex for drugs or money/divided by total # of participants) x 100
Time Frame: 1 year
Reporting Status: Not Posted

5. Secondary Outcome: The Percentage of Participants Who Report Sharing Injection Equipment
Description: (# participants reporting sharing injection equip/divided by total # of participants) x 100
Time Frame: 1 year
Reporting Status: Not Posted

6. Secondary Outcome: The Percentage of Participants With Household Incomes Below the Federal Poverty Level
Description: (# participants with incomes below federal poverty level/divided by total # of participants) x 100
Time Frame: 1 year
Reporting Status: Not Posted

7. Secondary Outcome: The Percentage of Opiate- and Cocaine-negative Urine Samples Post-intervention
Description: This will be measured after the intervention ends
Time Frame: Year 2
Reporting Status: Not Posted

8. Secondary Outcome: The Percentage of Participants Who Are Employed Post-intervention
Description: This will be measured after the intervention ends
Time Frame: Year 2
Reporting Status: Not Posted

9. Secondary Outcome: The Percentage of Participants Who Report Injecting Drugs Post-intervention
Description: This will be measured after the intervention ends
Time Frame: Year 2
Reporting Status: Not Posted

10. Secondary Outcome: The Percentage of Participants Who Report Trading Unprotected Sex for Drugs or Money Post-intervention
Description: This will be measured after the intervention ends
Time Frame: Year 2
Reporting Status: Not Posted

11. Secondary Outcome: The Percentage of Participants Who Report Sharing Injection Equipment Post-intervention
Description: This will be measured after the intervention ends
Time Frame: Year 2
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Cost-benefit of Treatment
Description: The Cost-Benefit Analysis (CBA) will compare the monetized benefits relative to costs
Time Frame: 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | IPS Only | IPS Plus Wage Supplement
All-Cause Mortality (participants affected / at risk) | 4/47 | 5/44
Serious Adverse Events (participants affected / at risk) | 8/47 | 5/44
Other Adverse Events (participants affected / at risk) | 11/47 | 8/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IPS Only (N=47) | IPS Plus Wage Supplement (N=44)
Death (General disorders) | 4 (4) | 5 (5)
leg amputated (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
kidney failure (Renal and urinary disorders) | 1 (1) | 0 (0)
stroke (Nervous system disorders) | 1 (1) | 0 (0)
upper respiratory problem (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IPS Only (N=47) | IPS Plus Wage Supplement (N=44)
chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
depression (Psychiatric disorders) | 2 (2) | 2 (2)
finger injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
flu-like symptoms (Gastrointestinal disorders) | 1 (1) | 0 (0)
hypertension (Cardiac disorders) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
psychiatric treatment (Psychiatric disorders) | 1 (1) | 1 (1)
foot pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
bumped eye (Eye disorders) | 0 (0) | 1 (1)
respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
seizure (Nervous system disorders) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-06): https://cdn.clinicaltrials.gov/large-docs/45/NCT02487745/Prot_SAP_000.pdf